CLINICAL TRIAL: NCT06740435
Title: Pilot Study Enhancing Telemedicine Care Delivery for Adults With Complex Type 2 Diabetes
Brief Title: Enhancing Telemedicine for T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Margaret Zupa, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY24060062; K23DK135794 (NIH)
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: Telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Telemedicine Care (Experimental): Specialty care for type 2 diabetes delivered via telemedicine by an endocrinologist, with additional multidisciplinary support from the diabetes care team.
  Interventions: Other: Enhanced Telemedicine for Type 2 Diabetes
- Usual Care (Active Comparator): Specialty care for type 2 diabetes delivered via telemedicine by an endocrinologist following usual clinical care protocols.
  Interventions: Other: Usual Telemedicine Endocrinology Care for T2D

INTERVENTIONS:
Other: Enhanced Telemedicine for Type 2 Diabetes — Telemedicine-based endocrinology specialty care for type 2 diabetes with multidisciplinary diabetes care team support including pre-visit preparation, in-visit support and self-management education, and post-visit follow-up.
  Arms: Enhanced Telemedicine Care
Other: Usual Telemedicine Endocrinology Care for T2D — Routine telemedicine-based endocrinology specialty care for type 2 diabetes, generally consisting of synchronous virtual visit with an endocrinologist and additional support including self-management education on an individualized basis.
  Arms: Usual Care

SUMMARY:
The goal of this pilot clinical trial is to assess feasibility of an intervention to deliver comprehensive, high-quality diabetes care through telemedicine among adults with type 2 diabetes who use insulin and have multiple chronic health conditions. The main question it aims to answer is:

Is an enhanced telemedicine intervention for type 2 diabetes compared to usual telemedicine care feasible?

Researchers will compare the enhanced telemedicine intervention to usual telemedicine care to see if there are differences in patient satisfaction or preliminary clinical outcomes.

Participants will complete 2-3 telemedicine diabetes care visits over approximately 6 months, as well as complete survey measures with each diabetes care visit. Patients in the intervention group will also receive additional support, including pre-visit preparation phone calls, diabetes self-management education and support aligned with their visits, and post-visit follow-up calls.

DETAILED DESCRIPTION:
This pilot study will compare an intervention to deliver high-quality diabetes care through telemedicine for adults with type 2 diabetes who have additional chronic health conditions and use insulin with usual telemedicine care. The investigators will assess feasibility, patient satisfaction, and preliminary clinical outcomes.

Fifty adults will be recruited from primary care practices. Once patients are confirmed eligible, they will be consented and enrolled. Patients will be randomized to the intervention arm or usual telemedicine care, stratified by age (above or below 65 years) and rurality, as these factors are associated with technological literacy and broadband access, which may impact telemedicine use and outcomes. Both groups will complete baseline survey measures and baseline clinical data will be collected via chart review. As this is a pragmatic pilot trial, intervention components will be delivered by usual clinical providers and staff for the intervention group. The telemedicine care intervention will include 2-3 synchronous visits with endocrinology providers over 6 months plus additional visits with multidisciplinary providers on an individualized basis. Telemedicine care will proceed as usual for the control group.

The investigators will focus pilot trial outcomes on standard metrics to assess feasibility for a future large trial. The investigators will also measure preliminary clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years or older
* Diagnosis of type 2 diabetes based on abbreviated ICD-10 code E11.X in medical record or self-report
* HbA1c greater than or equal to 8% based on most recent value at time of recruitment
* Patients must own or have access to a smart phone, tablet, or home computer with data or internet connection that allows access to video-based visits
* Patient must use insulin
* Patients must have >2 comorbid chronic health conditions
* Be able to provide informed consent
* Reside in Pennsylvania

Exclusion criteria:

* Age over 80 based on date of birth in electronic medical record
* Visit with an endocrinologist in the prior 1 years
* Dementia, ESRD, malignancy based on abbreviated ICD-10 codes below in medical record or self-report of associated condition

  * Dementia: A81.0x, F01.5x, F02.8x, F03.9x, F10.27, F10.97, F13.27, F13.97, F18.97, F19.17, F19.27, F19.97, G30.x, G31.0x, G31.1, G31.83, G31.85
  * Malignancy, except non-melanoma skin cancer: C00.x-C14.x, C15.x-C26.x, C3x.xx, C40.xx-C41.x, C43.x, C4A.xx, C45.x-C49.xx, C50.xxx, C51.x-C58, C60.x-C63.x, C64.x- C68.x, C69.xx-C72.x, C73-C76.x, C7A.xx, C80.xx-C96.x (except C90.x1, C91.x1, C92.x1, C93.x1, C94.x1, C95.x1)
  * ESRD N18.6
* Type 1, gestational, or other diabetes based on abbreviated ICD-10 codes below in medical record or self-report of associated condition

  * Type 1 diabetes: E10.X
  * Gestational diabetes: O24.X, E08.X
  * Other diabetes: E09.X, E13.2
* Pregnant or planning to become pregnant in next 6 months
* Currently enrolled in another diabetes management intervention study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment percentage | 12 months
  Percent of eligible patients approached who are enrolled
Loss to follow up | 6 months
  Percent of enrolled patients who do not complete study, defined as not completing at least 2 study visits and associated surveys

SECONDARY OUTCOMES:
Recruitment rate | 12 months
  Number of patients recruited per month
Eligibility percentage | 12 months
  Percent of patients approached who are eligible
Visit attendance | 6 months
  Percent of scheduled visits completed per patient
Number of between-visit contacts | 6 months
  Number of successful and attempted patient contacts by clinicians between visits per patient
Blood glucose data availability | 6 months
  Number of telemedicine visits with blood glucose data available at visit per patient
Patient satisfaction with telemedicine diabetes care | 6 months
  Percent of patients reporting satisfied or very satisfied on a 5-point Likert scale ranging from 1 "strongly disagree" to 5 "strongly agree" with the statement "Overall, I am satisfied with the quality of service being provided via telemedicine" with higher scores indicating greater satisfaction
Diabetes Treatment Satisfaction Questionnaire-static version | Baseline
  Total score of 8-item measure of global satisfaction with diabetes treatment regimen. The static version will be used at baseline. Items 1, 4, 5, 6, 7 & 8 are summed to produce a Treatment Satisfaction score (range:0 to 36). The higher the score, the greater the satisfaction with treatment. 'Perceived frequency of hyperglycaemia' (item 2) & 'Perceived frequency of hypoglycaemia' (item 3): Both rated: 6 ('most of the time') to 0 ('none of the time'). Here, lower scores indicate blood glucose levels closer to the ideal. Higher scores indicate problems.
Diabetes Treatment Satisfaction Questionnaire-change version | 6 months
  Total score of 8-item measure of global satisfaction with diabetes treatment regimen. The change version will be used at 6 months.Items 1, 4, 5, 6, 7 and 8 are summed to produce a Treatment Satisfaction (change) score (range: +18 to -18). The higher the score, the greater the improvement in satisfaction with treatment; the lower the score, the greater the deterioration in satisfaction with treatment. A score of 0 represents no change. Two remaining items ('Perceived change in frequency of hyperglycaemia' (item 2) and 'Perceived change in frequency of hypoglycaemia' (item 3)) are treated individually: Both rated: +3 ('much more of the time now') to -3 ('much less of the time now').
  Here, negative scores indicate fewer problems with blood glucose levels. Positive scores indicate more problems than before.
T2D Diabetes Distress Core Scale | Baseline and 6 months
  Change in total score of 8-item measure of diabetes-related distress over prior month from baseline to 6 months. The Diabetes Distress Core scale is scored by averaging the value for each item, ranked from 1 to 5 scale (score range 1-5), with higher scores indicating more distress.
HbA1c change | Baseline and 6 months
  Change in glycemic control from baseline to 6 months
Prescription of guideline-based GLP-1 receptor agonist | Baseline and 6 months
  Number of patients with indications for GLP-1 receptor agonist therapy who are prescribed the indicated medication
Prescription of guideline-based SGLT2 inhibitor | Baseline and 6 months
  Number of patients with indications for SGLT2 inhibitor therapy who are prescribed the indicated medication
Retinal examination | 6 months
  Number of patients with documentation of retinal examination performed in last year in medical record
Urine protein testing | 6 months
  Number of patients with documentation of urine protein testing performed in last year in medical record
Immunization-pneumococcal | 6 months
  Number of patients with documentation of pneumococcal vaccination in medical record
Immunization-influenza | 6 months
  Number of patients with documentation of influenza vaccination in medical record

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Zupa, MDMS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset including limited demographic, encounter, laboratory result, clinical observations, medication orders, care utilization, and survey (intervention satisfaction, treatment satisfaction, diabetes distress) data will be created. To protect research participant identities, datasets will not include any potentially identifying participant information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available no later than 12 months and ending 36 months after the primary trial results are published.
Access Criteria: No access will be granted until the requesting investigator vetting process is completed including an IRB-approved protocol and data use agreement with the University of Pittsburgh.The data that may be shared includes: de-identified participant data, tables, figures, appendices, analysis plan, and protocol.